CLINICAL TRIAL: NCT03926663
Title: Effects of Intranasal Injection of Dexmedetomidine Plus Bupivacaine on Anesthesia & Analgesia in Septoplasty Surgeries
Brief Title: Intranasal Injection of Dexmedetomidine and Bupivacaine in Septoplasty Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Zayed, Lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FMBSUREC/05032019/Moselhy
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Intranasal Dexmedetomidine; Intranasal Bupivacaine; Septoplasty Surgeries
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group Bupivacaine (Experimental): Group B; will receive 0.25% bupivacaine (with an average dose of 1-1.5 mg/kg) as preincisional local infiltration of the nasal mucosa of the nasal septum ,injected once before surgical intervention
  Interventions: Drug: Bupivacaine
- group Bupivacaine +Dexmedetomidine (Active Comparator): group B+D; will receive 0.25% bupivacaine (with an average dose of 1-1.5 mg/kg) + 0.2 μg/kg dexmedetomidine preincisional local infiltration of the nasal mucosa of the nasal septum,injected once before surgical intervention.
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine, a potent α-2 adrenoceptor agonist, is approximately 8 times more selective toward the α-2 adrenoceptors than clonidine.
  Patients will receive 0.25% bupivacaine (with an average dose of 1-1.5 mg/kg) + 0.2 μg/kg dexmedetomidine preincisional local infiltration of the nasal mucosa.
  Other Names: Precedex,
  Arms: group Bupivacaine +Dexmedetomidine
Drug: Bupivacaine — patients will receive 0.25% bupivacaine (with an average dose of 1-1.5 mg/kg) preincisional local infiltration of the nasal mucosa.
  Other Names: Marcaine

SUMMARY:
Pain is particularly common after nasal surgery, especially when bone manipulation and periosteal irritation are involved. Appropriate pain control is an important consideration in the post-surgical management of patients.

DETAILED DESCRIPTION:
Multiple researches and clinical observations suggest that pain reduction can be achieved in nasal surgery by using local anesthesia.The combination of local anesthetic infiltration, directly in the surgical field, with general anesthesia provides beneficial analgesic effects by blocking nociceptive pathways, and there by it reduces the need for systemic analgesics.

The use of α-2 Adrenergic receptor (adrenoceptor) agonists in anesthesia were the focus of interest for their sedative, analgesic, and perioperative sympatholytic and cardiovascular stabilizing effects with reduced anesthetic requirements. α-2 agonists, inhibit substance P release in the nociceptive pathway at the level of the dorsal root neuron; in addition, α-2 adrenergic receptors located at nerve endings may have a role in the analgesic effect of the drug by preventing norepinephrine release.

In this study, the combined effects of dexmedetomidine with bupivacaine as local anesthetics vs bupivacaine, will be investigated in septoplasty to determine the need for rescue drugs as propanlol and nitroglycerine, as hypotensive agents,for bloodless surgical field and optimal procedure for pain control

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18- 60 years
* ASA physical status I
* Undergoing septoplasty

Exclusion Criteria:

* Patients with cardiovascular disease (congestive heart failure, coronary artery disease, hypertension.
* History of renal or hepatic insufficiency
* Endocrinal Diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The precentage of patients that will take rescue drugs as nitroglycerin, propranolol. | 3 hours
  the number of patients that will need rescue drugs: propranolol 1mg will be given then after 15 minutes (with no improvement of the surgical field) nitroglycerin (NTG) infusion will be added in a titrated manner 0.1-0.5 μg/kg/min gradually till the target MAP (±60 mmHg) is reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine,Beni-Suef University, Banī Suwayf, Egypt